CLINICAL TRIAL: NCT00619788
Title: Prospective, Multicenter, Non-randomized Clinical Trial Investigating the Safety and Efficacy of the AngioSculpt Scoring Balloon Catheter (AngioScore, Inc.) for the Treatment of Femoropopliteal Stenotic Disease.
Brief Title: FeMoropopliteal AngioSculpt™ SCoring BallOon CaTheter Study
Acronym: MASCOT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Collaborators: AngioScore, Inc. (Industry)
Responsible Party: Flanders Medical Research Program, Flanders Medical Research Program
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-003
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients receiving 4.0-5.0mm AngioSculpt Scoring Balloon Catheter (AngioScore, Inc.) for femoropopliteal use
  Interventions: Device: 4.0-5.0mm AngioSculpt Scoring Balloon Catheter

INTERVENTIONS:
Device: 4.0-5.0mm AngioSculpt Scoring Balloon Catheter — The AngioSculpt Scoring Balloon Catheter is a line of innovative angioplasty catheters comprising an angioplasty balloon surrounded by a unique system of nitinol scoring elements. Creating focal concentrations of dilating force, the scoring elements score arterial lesions as the balloon expands.

SUMMARY:
This investigation is designed to demonstrate the efficacy and safety of the 4.0-5.0mm AngioSculpt Scoring Balloon Catheter (AngioScore, Inc.) for femoropopliteal use in a controlled clinical investigation.

The scoring balloon is a semi-compliant balloon encircled by 3 spiral struts with a nitinol scoring element, which theoretically provides targeted scoring of lesions, by concentrating the dilation force thus minimizing barotrauma, elastic recoil and uncontrolled dissection. This may improve the outcome of the intervention and reduce the number of stents required.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic (>50%) or occlusive atherosclerotic disease of the femoropopliteal arteries (primarily superficial femoral arteries - SFA)
* Length of lesion >5 cm or 2 times the AngioSculpt balloon length (whichever is longer)
* Reference vessel diameter should be 4.0-6.0 mm
* Life altering claudication or critical limb ischemia (Rutherford 3-5)
* No untreated inflow-limiting arterial lesions
* At least single vessel run-off until the ankle
* The patient must be > 18 years.
* Life-expectancy of more than 12 months
* The subject or legal guardian has been informed of the nature of the evaluation; agrees to its provisions and has signed informed consent
* The patient is capable to follow all evaluation requirements.

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for available catheter design
* Length of lesion is ≥5 cm or requires more than two overlapping AngioSculpt balloon inflations (whichever is longer) to cover the entire lesion (however, more than two inflations are permitted within an acceptable lesion length)
* The patient has a known allergy to heparin, aspirin or other anticoagulant/antiplatelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies
* The patient has a history of prior life-threatening contrast media reaction
* The patient is currently enrolled in another investigational device or drug trial
* The patient is currently breast-feeding, pregnant or intends to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Complication Free Survival at 1 month post-procedure (complications = major amputations defined as amputations at or above the ankle, any cause of death and TLR) | 1 month

SECONDARY OUTCOMES:
patency of the target lesion. Primary patency is defined as the absence of: a) target lesion revascularization (TLR); b) major amputation due to lesion restenosis or occlusion; c) conversion to bypass surgery and d) untreated significant stenosis on CFDU | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Peeters, MD, Principal Investigator — Imelda Hospital, Bonheiden, Belgium
Locations (3):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ St-Blasius, Dendermonde
- Herzzentrum, Leipzig, Germany